CLINICAL TRIAL: NCT02134717
Title: An Interventional Study of the Effect of CCR5 Inhibition With Maraviroc on Immune Cells in the the Lung and in Peripheral Blood of Patients With Sarcoidosis
Brief Title: Impact of Chemokine Receptor 5 (CCR5) Inhibition on Sarcoidosis Immunophenotypes
Acronym: GRADS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor recruitment
Sponsor: Kevin F. Gibson (Other)
Collaborators: University of Pittsburgh (Other)
Responsible Party: Sponsor-Investigator, Kevin F. Gibson, MD, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: U01HL112711 (NIH)
Record Dates: First submitted 2014-04-30; First posted 2014-05-09 (Estimated); Results first posted 2017-07-18 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Sarcoidosis
Keywords: sarcoidosis; CCR5 inhibition; maraviroc
MeSH Terms: conditions — Sarcoidosis | interventions — Maraviroc; Bronchoalveolar Lavage; Phlebotomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- sarcoidosis stage II (Experimental): All subjects with active stage II sarcoidosis with or without skin disease will receive the drug maraviroc 300mg to be taken orally twice a day for 6 weeks duration.
  Interventions: Drug: all subjects will receive maraviroc 300mg orally twice a day for 6 weeks; Procedure: Bronchoscopy with bronchoalveolar lavage; Procedure: venipunctures; Procedure: Skin biopsy

INTERVENTIONS:
Drug: all subjects will receive maraviroc 300mg orally twice a day for 6 weeks
  Other Names: maraviroc; selzentry
Procedure: Bronchoscopy with bronchoalveolar lavage — Bronchoscopy employs a flexible instrument that is inserted into the trachea and proximal airways after topical anesthesia. Bronchoalveolar lavage involves the instillation of saline solution through the bronchoscope into the airways followed by recovery under suction to collects lung fluid containing cells and proteins.
Procedure: venipunctures — Venipunctures will be performed at study entry, after two weeks, and at the end of the study to collect blood for research studies and safety laboratories.
Procedure: Skin biopsy — For subjects with sarcoidosis skin lesions, an optional skin biopsy specimen may be collected for research studies.

SUMMARY:
The study hypothesizes that inhibition of the receptor CCR5 by maraviroc will diminish inflammation in patients with sarcoidosis. Subjects with active sarcoidosis will first undergo bronchoscopy with bronchoalveolar lavage to recover lung immune cells for baseline analysis. They will then receive the drug maraviroc for 6 weeks duration. They will then undergo a repeat bronchoscopy with bronchoalveolar lavage to recover lung immune cells for analysis following maraviroc treatment.

DETAILED DESCRIPTION:
The investigators hypothesize that inhibition of CCR5 by maraviroc may have a beneficial immunomodulatory effect on the granulomatous inflammation of pulmonary sarcoidosis. The specific aim of this proposal is the investigate the effect of CCR5 inhibition on the trafficking of mononuclear cells to the lung, skin, peripheral blood in subjects with active sarcoidosis exposed to the CCR5 inhibitor, maraviroc. A second aim will be to isolate by cell sorting cluster of differentiation 4 (CD4)+CCR5+ T cells for amplified gene expression profiling before and after CCR5 inhibition, experiments the investigators believe will elucidate genes associated with downstream activation and inhibition of CCR5 receptor function.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven sarcoidosis from any site (noncaseating granulomas without other causes).
2. Diagnosis of active sarcoidosis (Sec. 5.5.4.t) clinical stage II by Chest X-ray (CXR).
3. Forced Vital Capacity (FVC) >45% and Diffusing Capacity for Carbon Monoxide (DLCO) >50% of predicted values.
4. Evidence of active sarcoidosis (see criteria above)
5. Able and willing to complete all study procedures (e.g., bronchoscopy, post-drug surveillance)
6. Age: 18+ years old (prevalence greatest in young adults; pediatric maraviroc safety not established).
7. Not on immunosuppression for sarcoidosis at the time of recruitment, (e.g., steroids, tumor necrosis factor alpha (TNF-a) blockade)
8. Liver function (transaminases, bilirubin), coagulation (International Normalized Ratio (INR), partial thromboplastin time (PTT), platelet count), blood urea nitrogen (BUN), creatinine, and white blood count (WBC) within normal limits.
9. If female: negative pregnancy test, agreement to use reliable contraception if of childbearing potential 30 days prior and for 30 days after study completion (drug safety during pregnancy not established).
10. Negative HIV and HBsAg tests

Exclusion Criteria:

1. Diagnosis of infection based upon clinical evaluation and/or microbial testing.
2. The diagnosis of any disease involving the heart, lungs, liver (HVC), kidney, hematologic, endocrine, or Gl systems which, in the judgment of the PI, would pose an undue risk to the subject if they participated in this study. This includes but is not limited to diabetes, uncontrolled hypertension, liver disease (HVC), or history of malignancy.
3. Medications that will either inhibit or induce CYP3A4 (including St John's Wort)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2014-01; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin F Gibson, MD, Principal Investigator — DorothyP. and Richard P. SImmons Center for Interstitial Lung Disease at the University of Pittsburgh
Locations (1):
- Dorothy P. and Richard P. Simmons center for Interstitial lung Disease at the University of Pittsburgh, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects with sarcoidosis stage II and active disease
Pre-assignment Details: Willing to undergo two Bronchoalveolar lavages
Groups:
- Sarcoidosis Stage II: All subjects with active stage II sarcoidosis with or without skin disease will receive the drug maraviroc 300mg to be taken orally twice a day for 6 weeks duration.
  all subjects will receive maraviroc 300mg orally twice a day for 6 weeks
  Bronchoscopy with bronchoalveolar lavage: Bronchoscopy employs a flexible instrument that is inserted into the trachea and proximal airways after topical anesthesia. Bronchoalveolar lavage involves the instillation of saline solution through the bronchoscope into the airways followed by recovery under suction to collects lung fluid containing cells and proteins.
  venipunctures: Venipunctures will be performed at study entry, after two weeks, and at the end of the study to collect blood for research studies and safety laboratories.
  Skin biopsy: For subjects with sarcoidosis skin lesions, an optional skin biopsy specimen may be collected for research studies.
Period: Overall Study
Arm/Group | Sarcoidosis Stage II
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: This study was terminated due to inadequate funding to complete the recruitment and analysis.
Arm/Group | Sarcoidosis Stage II
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants] — This study was terminated due to inadequate funding to complete the recruitment and analysis. Population: This study was terminated due to inadequate funding to complete the recruitment and analysis.
  Participants
    <=18 years | 0
    Between 18 and 65 years | 3
    >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] — Population: This study was terminated due to inadequate funding to complete the recruitment and analysis.
  years | 37 [23 to 58]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 1
Region of Enrollment [Number; unit: participants] — Population: This study was terminated due to inadequate funding to complete the recruitment and analysis.
  participants
    United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Total Cell Count and Differentials in Blood and Bronchoalveolar Lavage Fluid Pre- and Post Maraviroc
Description: General indicators of inflammation following chemokine receptor 5 (CCR5) inhibition in blood and bronchoalveolar lavage
Time Frame: 6 weeks
Population: Data could not be analyzed
Arm/Group | Sarcoidosis Stage II
Number analyzed (Participants) | 0

2. Secondary Outcome: Mononuclear Cell (MNC) Activation and T-cell Differentiation
Description: MNC activation and T-cell differentiation before and after CCR5 inhibition.
Time Frame: 6 weeks
Population: Study was terminated before data were collected for this outcome measure.
Arm/Group | Sarcoidosis Stage II
Number analyzed (Participants) | 0

3. Secondary Outcome: Chemokine Receptor 5 (CCR5) Expression Among These Immune Effector Cells
Description: CCR5 expression among these immune effector cells before and after CCR5 inhibition.
Time Frame: 6 weeks
Population: Study was terminated before data were collected for this outcome measure.
Arm/Group | Sarcoidosis Stage II
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Sarcoidosis Stage II
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 0/3

LIMITATIONS AND CAVEATS:
This study was terminated due to inadequate funding to complete the recruitment and analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No